CLINICAL TRIAL: NCT01682096
Title: Usefulness of Coronary CTA for the Diagnosis of Acute Coronary Syndrome in the Emergency Room.
Brief Title: Pilot Safety Study of Coronary CTA for the Diagnosis of Acute Coronary Syndrome in the Emergency Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José Ortiz (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, José Ortiz, MD, PhD,, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI09/90513
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease; Cardiac Death; Myocardial Infarction
Keywords: Chest pain; Emergency room; Acute coronary syndrome; Computed tomography coronary angiography; Stress echocardiography
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Death; Myocardial Infarction; Chest Pain; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computed coronary angiography (CTA) (Active Comparator): Patients will undergo a MDCT as the initial diagnostic test to rule out Acute Coronary Syndrome
  Interventions: Radiation: computed coronary angiography
- Exercise stress echocardiography (Active Comparator): Patients will undergo exercise stress echocardiography as the initial diagnostic test to rule out acute coronary syndrome.
  Interventions: Procedure: Exercise stress echocardiography

INTERVENTIONS:
Radiation: computed coronary angiography — Patients will be pre-medicated with atenolol 50 mg 1h prior to the scan.
  Other Names: coronary cta; SIEMENS 64/128 slice CT scanner
  Arms: Computed coronary angiography (CTA)
Procedure: Exercise stress echocardiography — Limited by symptoms
  Other Names: Treadmil exercise stress echocardiography
  Arms: Exercise stress echocardiography

SUMMARY:
The Diagnosis of acute coronary syndrome in patients presenting with acute chest pain is problematic when both, electrocardiogram and serum troponins are normal. Multidetector row computed tomography angiography (CTA) allows direct and rapid non-invasive visualization of coronary artery disease.

The investigator's aim is to assess the diagnostic accuracy and safety of a novel diagnostic strategy based on MDCT as compared to a strategy using stress echocardiography in the workup of patient with chest pain, normal electrocardiogram, normal troponins and suspected coronary artery disease. Additionally, the cost associated with both strategies will be compared.

Methods. A total of 150 patients with acute chest pain coming to the emergency room with intermediate probability of significant coronary artery disease, normal ECG and troponins will be prospectively randomized to MDCT or stress echocardiography with exercise. Patients showing coronary stenosis >50% at MDCT or abnormal stress echocardiography or inconclusive results will be admitted for further study. The primary endpoint of the study is the detection of an acute coronary syndrome, defined as typical or atypical angina with documented significant coronary artery disease (>50% stenosis) on invasive coronariography, a positive stress test or the occurrence of cardiac death, myocardial infarction or need for revascularization during 6 month follow-up. All MDCT angiograms and echocardiograms will be evaluated by an experienced radiologist and cardiologist.

DETAILED DESCRIPTION:
Design and Aim: This is a prospective pilot study to evaluate the role of multidetector row computed tomography angiography (CTA) to rule out Acute Coronary Syndrome among patients presenting to the ER with chest pain complaints, non-diagnostic ECG and normal troponins and intermediate pre-test probability for significant CAD.

Methods: Following the initial clinical evaluation and the results of initial ECG, blood test and X-ray, patients meeting the inclusion criteria will be randomized to undergo either a CTA scan or a Exercise Stress Echocardiogram to rule out significant coronary artery disease.

CTA will be carried out in a 64 or 128 slice-CT Scanner (SIEMENS,Somaton Sensation 64 or 128-Flash Definition)following iv administration of iodinated contrast (bolus: 5cc x acquisition time (seg)+ 10 cc). Images will be interpreted by two experienced physicians (radiologist and cardiologist)

Stress Echocardiography will be performed and interpreted by an experienced Echocardiographer (cardiologist).

Clinical decision making: Patients with a positive or inconclusive test in each arm will be admitted to the hospital for treatment or further additional testing, while patients with negative results will be discharged from the ER.

Safety issues: A phone call and chart review will be performed one month and 6 months follow-up to register the occurrence of any major adverse cardiac events, as well as new consultation for chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient is in Sinus Rhythm
* Typical or atypical chest pain lasting more than 5 min in the last 24 hs.
* Estimated pre-test probability of significant coronary artery disease more than 15%.
* Absence of ECG changes suggestive of myocardial ischemia (ST-segment deviation >1 mm or T Wave inversion > 4 mm in at least two contiguous leads).
* Negative initial troponins I at admission (<0.05 ng/ml)

Exclusion Criteria:

* Known allergy to iodinated contrast.
* Known renal insufficiency or Creatinine >1.5 mg/dl at admission.
* History of known coronary artery disease or prior myocardial revascularization
* Any of the following:hemodynamic instability, persistent chest pain despite treatment, Systolic blood pressure <100 mm Hg.
* Cardiac arrhythmia with rapid or irregular ventricular response.
* Inability to perform an exercise test.
* Patient is incapable of providing informed consent.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Acute Coronary Syndrome during admission or occurrence of Major Acute Cardiac Events after discharge | 6 months
  Major adverse cardiac events include: All cause mortality, acute myocardial infarction, need for coronary revascularization

SECONDARY OUTCOMES:
Major adverse cardiac events on follow-up | 6 months
  Safety endpoint: occurrence of MACE among discharged patients in whom acute coronary syndrome has been ruled out according to the test results
Costs during admission (Euros) | 6 months
  The total costs derivated from the admission between the two arms of the study will be compared. Results will be reported in Euros, and will include the costs of the CTA or Stress echocardiography as well as additional tests performed during admission.

OTHER OUTCOMES:
Time to clinical decision | first 24 hs.
  Time from patient admission to the clinical decision (admission for further testing or discharge from the ER) between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: José T Ortiz-Perez, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain